CLINICAL TRIAL: NCT01327092
Title: Injury Prevention in a Home Visitation Population
Brief Title: Cincinnati Home Injury Prevention Study
Acronym: CHIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Dr. Kieran Phelan, Principal Investigator, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R01HD066115-01A1 (NIH)
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Injury in the Home
Keywords: Injury; Injury Prevention; Cincinnati Home Injury Prevention; Injury Hazards; Modifiable Injury Hazards; CHIP; Literacy Promotion; Reduce exposure to injury hazards; preventable and medically attended injury; young children
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Literacy Group (No Intervention): Families in the Literacy Group (control group)will receive a program which seeks to promote literacy by providing developmentally appropriate books and other reading-related materials to children and encouraging mothers to develop an interest in reading with their child. After enrollment and randomization, CHIP staff will visit these control group homes, assess the mother's interest in and barriers to reading with her child, council mothers about the importance of literacy and reading books to their child, and children will be given age appropriate books and other materials to promote literacy.
- Injury Intervention Group (Experimental): Injury Intervention Group: In homes of children who are randomized to the injury intervention arm of the trial, a comprehensive survey of injury hazards in living spaces will be undertaken. In addition to quantifying hazards, the area of living spaces will be obtained to allow the determination of both the number and density (number of hazards per 100 sq ft) of injury hazards. If one or more injury hazards are identified, they will be removed and/or modified to reduce exposure and injury risk. The intervention is focused on areas in living spaces below 1 meter (~39 inches) in height from (the 75th percentile in height or eye-level for a 3-year old US male toddler) which might be easily reached or climbed on by children less than 4 years
  Interventions: Other: Injury Intervention Group

INTERVENTIONS:
Other: Injury Intervention Group — The hazards identified in the home will be reviewed with the parent and the proposed interventions will be presented. Intervention options are designed and prioritized so that the most passive and durable interventions are recommended first (e.g. self-closing, self-locking stair gate) and progressively less 'passive' and less durable options last (e.g. area gate, pressure mounted gate, or refusal of intervention).
  Arms: Injury Intervention Group

SUMMARY:
One aim of this study is to test the efficacy of the installation of multiple, passive measures to reduce exposure to injury hazards in the homes of young children of first-time mothers and reduce childhood injury. The study also seeks to identify sub-groups of mothers and children who benefit most from the intervention and examine the potential moderating effect of maternal depressive symptoms, the intensity of supervisory behavior, and child temperament and activity, on the intervention and subsequent injury outcomes.

Specific Aim 1 Hypotheses:

H1.1: The housing units randomly assigned to the intervention group will have a significant decrease in the number and density (number per area) of residential injury-related hazards compared with control group units.

H1.2: Children who are randomized to the intervention group (e.g. installation of multiple, passive measures to reduce exposure to residential injury hazards) will have a 50% reduction in modifiable and medically-attended injuries compared with children in the control group followed-up for 24-months in intention-to-treat analyses.

Specific Aim 2: Hypotheses H2.1: Persistent maternal depressive symptoms will moderate the effects of the intervention on childhood injury in the home; households and children of mothers with higher levels of symptoms will have more hazards and injuries.

H2.2: Children of mothers with less intense maternal supervisory behavior over the course of the intervention follow-up will have higher rates of injury.

H2.3: Children scoring high in activity on the Carey Temperament Scale will experience reduced benefits of the intervention on childhood injury in the home.

DETAILED DESCRIPTION:
Injury remains the leading cause of morbidity and mortality for U.S. children after the first year of life and the home is the leading location of injury for younger U.S. children. Residential injury results in more than 1.7 million emergency visits in children younger than 5 years of age annually in the U.S. resulting in over $3 billion in medical care costs and $800 per emergency visit. Therefore, interventions that can effect sizable reductions in childhood injury in the home could result in substantial reductions in pain and suffering while saving potentially hundreds of millions of dollars in healthcare costs.

Previous trials have failed to achieve comprehensive and durable installation of home safety products to reduce exposure to injury hazards in the indoor environments of young children. Children of mothers who are eligible and enrolled in home visitation programs and children of mothers with elevated depressive symptoms have been shown to be at risk for injury in the home. Inadequate maternal supervisory behavior has also been shown to increase the risk for home injury. This project will test the efficacy of an intervention to reduce exposure to injury hazards in the home and subsequent preventable and medically attended injury in young children of first-time, impoverished mothers.

This randomized control trial will test the efficacy of a public health intervention to reduce exposure to injury hazards through the proper installation of safety devices in the home and subsequent preventable and medically attended injury in the Every Child Succeeds (ECS) population. Participants will be randomized to either receive injury prevention measures or be a part of a literacy effort that provides developmentally appropriate books and reading materials to mothers and children, and encourages mothers to gain interest in reading with their child.

Mothers that participate in the Every Child Succeeds (ECS) home visitation program, have completed at least one ECS home visit, and have a child less than 5 months of age will be enrolled in the study. Index children will be followed for 24 months after randomization and interventions or up to the age of approximately 36 months. Measures of maternal and child psychology, child behavior and temperament will be obtained during home visits. Maternal supervision and childhood injuries will be assessed repeatedly during quarterly phone questionnaires and home visits.

Experimental Group: In homes of children randomized to the intervention arm of the trial, a comprehensive observational survey of living spaces will be undertaken. The study will examine living spaces to which a child may be exposed including 5 high-exposure, high-risk areas (main activity room, kitchen, child's bedroom and bathrooms, and stairways). In addition to quantifying hazards, the area of rooms will be obtained allowing for determination of both the number and density of injury hazards.

The hazards identified by the intervention team will be reviewed with the parent and the proposed interventions will be presented. Intervention options are designed and prioritized so that the most passive and durable interventions are recommended first and progressively less 'passive' and less durable options last. After consent is obtained, passive measures will be installed across the living space as indicated.

One goal of the study is to determine whether installed products that modify exposure to the injury hazards can reduce unintentional injury across the leading mechanisms for young children over time. Another goal is to determine the required maintenance of installed products over time. At routine home visits or at the request of a participant prior to the 18-month follow-up time point, installed interventions will be assessed for their presence and function and broken or malfunctioning products will be repaired or replaced if it is within the study budget. Additionally, if the study budget allows, the investigators will repeat the injury hazard survey and perform the installation intervention if a family relocates prior to the child being 24-months of age, within a 3 hour driving radius of CCHMC, and has not moved more than three times.

Control Group: Mothers and children randomly assigned to the control condition will also benefit from participation in the trial. Similar to the intervention arm, they will undergo home surveys and annual visits for assessment of injury hazards. In addition, families in this control group will receive a program which seeks to promote literacy by providing developmentally appropriate books, materials and possibly a library card to children and encouraging mothers to develop an interest in reading with their child. After enrollment and randomization, CHIP staff will visit these control group homes, assess the mother's interest in and barriers to reading with her child, and council mothers about the importance of literacy and reading books to their child.

ELIGIBILITY:
Inclusion:

* Mothers enrolled in the ECS program who have completed at least one ECS home visit

Exclusion- Mothers who:

* Have a child greater than 5 months of age
* Are non-English speaking
* Live beyond a 3-hr driving radius
* Have plans to relocate outside of a 3-hour driving radius from Cincinnati Children's Hospital in the next 12 months at the time of screening
* Mothers with ECS accounts marked as "Other" such as HMG Part C (having a chronic illness, congenital disorder or developmental delay), HMG At-Risk, first time fathers in Kentucky, etc.
* index child is a twin

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2010-09; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Any modifiable and medically-attended injury in enrolled children | Quarterly (baseline & annual home visits, quarterly phone surveys) (up to 4 years)
  Primary outcome measures will include any phone calls, clinic, and ED visits for falls, cuts/lacerations, contusion/crush, burn/scald, abrasions, and poisoning injuries sustained by enrolled children in the home that were potentially modifiable by the installed safety products. Modifiable injury events are defined as those whose hazard exposure and associated mechanism was potentially modified by the intervention (ie stairgate reducing exposure to a stairway and subsequent stairway fall injury) and include fall, cut/pierce, struck/strike, burn, and poisoning mechanisms.

SECONDARY OUTCOMES:
Correlation of self-reports of non-emergent but medically attended residential injuries in enrolled children. | Annually (up to 4 years)
  Verification of self-reports will be accomplished through annual medical record review. Emergency visit reports will be confirmed by matching the maternal report to the Hamilton County Injury Surveillance System (HCISS) a data repository of all injuries resulting in emergency visits, hospitalizations, and deaths for all persons presenting to Hamilton County hospitals and emergency departments.

CONTACTS AND LOCATIONS:
Overall Officials: Kieran Phelan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Phelan KJ, Khoury J, Xu Y, Lanphear B. Validation of a HOME Injury Survey. Inj Prev. 2009 Oct;15(5):300-6. doi: 10.1136/ip.2008.020958. PMID 19805597